CLINICAL TRIAL: NCT01767714
Title: A Phase 3 Multicenter, Randomized, Double-Blind, Placebo-Controlled, Comparative Trial of Plerixafor (0.24 mg/kg) Plus G CSF (10 µg/kg) Versus G CSF (10 µg/kg) Plus Placebo to Mobilize and Collect ≥5 × 106 CD34+ Cells/kg in Non-Hodgkin's Lymphoma (NHL) Patients for Autologous Transplantation
Brief Title: Evaluation of Plerixafor Plus G-CSF to Mobilize and Collect 5×10^6CD34+ Cells/kg in Non-Hodgkin's Lymphoma (NHL) Patients for Autologous Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC12482; MOZ14409 (Other: Genzyme); U1111-1131-0145 (Other: UTN)
Record Dates: First submitted 2012-12-17; First posted 2013-01-14 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: hematopoietic stem cell transplantation
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Granulocyte Colony-Stimulating Factor; Granisetron; Filgrastim; plerixafor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- G-CSF + plerixafor (Experimental): Patients will receive G-CSF for 4 mornings for mobilization, followed by another dose each morning before apheresis on days that the patient is to continue apheresis (up to 8 doses total). Patients will also receive plerixafor in the evening up to a maximum of 4 doses.
  Interventions: Drug: Granulocyte-colony stimulating factor (G-CSF); Drug: Plerixafor
- G-CSF + Placebo (Placebo Comparator): Patients will receive G-CSF for 4 mornings for mobilization, followed by another dose each morning before apheresis on days that the patient is to continue apheresis (up to 8 doses total). Patients will also receive placebo in the evening up to a maximum of 4 doses.
  Interventions: Drug: Granulocyte-colony stimulating factor (G-CSF); Drug: Placebo

INTERVENTIONS:
Drug: Granulocyte-colony stimulating factor (G-CSF) — 10 µg/kg/day G-CSF, administered by subcutaneous (SC) injection
  Other Names: GRAN®, Filgrastim
Drug: Plerixafor — 0.24 mg/kg/day subcutaneous injection
  Other Names: Mozobil, AMD3100, GZ316455
  Arms: G-CSF + plerixafor
Drug: Placebo — 0.24mg/kg/day placebo (0.9% Sodium Chloride) administered by subcutaneous injection
  Arms: G-CSF + Placebo

SUMMARY:
The study is to determine if NHL patients mobilized with G-CSF (10 µg/kg/day [GRAN® only]) plus 0.24 mg/kg/day of plerixafor are more likely to achieve a target number of ≥5 × 10^6 CD34+ cells/kg in 4 or fewer days of apheresis than NHL patients mobilized with G-CSF plus placebo.

DETAILED DESCRIPTION:
Eligible patients who are unable to achieve adequate apheresis cell counts may enter an Open-Label Rescue Period where they will receive plerixafor, following the same study schedule as during the Double-Blind Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

* Has a biopsy-confirmed diagnosis of NHL
* Is in first or second complete remission or partial remission, defined for the purpose of this study as complete or partial response following first- or second-line therapy
* Treatment with an autologous peripheral HSC transplant is planned and the patient is eligible for autologous transplantation
* Has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Has recovered from all acute toxic effects of prior chemotherapy or other cancer treatment.
* Has an actual body weight <175% of their ideal body weight (IBW)
* The patient agrees to use a highly effective method of contraception from Day 1 through ≥3 months following plerixafor treatment.

Exclusion Criteria:

* Concurrent serious illness and pathological conditions
* Has undergone previous HSC collections or collection attempt
* Has had any autologous or allogeneic HSC transplant
* Has active central nervous system (CNS) involvement
* Bone marrow lymphoma cells involvement >20%, as assessed by bone marrow biopsy within 4 months before signing the ICF
* Has received radiation therapy to the pelvis
* Has a diagnosis of all leukemias including any type of CLL
* Active infection
* Pregnant or nursing
* Anticipated post-transplant chemotherapy and/or radiation therapy below the diaphragm
* Received any prior radio-immunotherapy
* Prior 1,3-bis(2-chloroethyl)-1-nitroso-urea (BCNU) within 6 weeks prior to first dose of G-CSF
* Prior cancer therapy, other investigational therapy within 4 weeks prior to first dose of G-CSF
* Prior granulocyte/macrophage-colony stimulating factor (GM-CSF) or pegfilgrastim within 3 weeks prior to the first dose of G-CSF
* Prior G-CSF within 2 weeks prior to the first dose of G-CSF
* Inadequate organ funtion evidenced by unacceptable laboratory result

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of patients who meet the target of ≥5 × 10^6 CD34+ cells/kg in 4 or fewer days of apheresis | Days 5- Day8

SECONDARY OUTCOMES:
Number of patients who achieve ≥2 × 10^6 CD34+ cells/kg within 4 or fewer days of apheresis | Day 5 - Day 8
Number of days of apheresis to collect ≥2 × 10^6 CD34+ cells/kg | Up to achieve the target of collecting ≥2 × 10^6 CD34+ cells/kg
Number of days of apheresis to collect ≥5 × 10^6 CD34+ cells/kg | Up to achieve the target of collecting ≥5 × 10^6 CD34+ cells/kg
Total number of CD34+ cells collected | Day 5 - Day 8
Time from transplantation to neutrophil and platelet (PLT) engraftment | up to 30 days post-transplantation
Number of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | from signed Informed Consent Form (ICF) to 30 days post-transplant and then ongoing as needed
Maximum plasma concentration (Cmax) | Day 4 - Day 5
Time to reach Cmax (Tmax) | Day 4 - Day 5
Area Under the Curve 0 to 10 hours post-dose (AUC0-10) | Day 4 - Day 5
Area Under the Curve 0 to last observed concentration (AUClast) | Day 4 - Day 5
Area Under the Curve (AUC) | Day 4 - Day 5
Percentage of extrapolation of AUC (AUCext) | Day 4 - Day 5
Half life (T1/2) | Day 4 - Day 5
Volume of distribution (Vz/F) | Day 4 - Day 5
Total body clearance (CL/F) | Day 4 - Day 5
Peripheral blood CD34+ cell counts (Pharmacodynamic analysis) | Day 4 - Day 5
The fold-increase in the number of circulating CD34+ following the first dose of plerixafor or placebo, with the first apheresis day (Day 5) value serving as the primary estimate | Day 5 - Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (16):
- China (16):
  - Investigational Site Number 156017, Beijing
  - Investigational Site Number 156001, Beijing
  - Investigational Site Number 156005, Beijing
  - Investigational Site Number 156002, Beijing
  - Investigational Site Number 156003, Beijing
  - Investigational Site Number 156020, Chongqing
  - Investigational Site Number 156016, Fuzhou
  - Investigational Site Number 156021, Guangzhou
  - Investigational Site Number 156011, Hangzhou
  - Investigational Site Number 156018, Nanjing
  - Investigational Site Number 156009, Shanghai
  - Investigational Site Number 156010, Suzhou
  - Investigational Site Number 156008, Tianjin
  - Investigational Site Number 156013, Wuhan
  - Investigational Site Number 156015, Xi'an
  - Investigational Site Number 156022, Zhengzhou